CLINICAL TRIAL: NCT03451721
Title: Observation of ImageReady™ MR Conditional Defibrillation System in China (MR ICD)
Brief Title: Observation of ImageReady™ MR Conditional Defibrillation System in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C2082
Record Dates: First submitted 2017-09-04; First posted 2018-03-02 (Actual); Results first posted 2020-04-24 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2019-09

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ImageReady™ MR Conditional Defibrillation System (Experimental): 1. Subject is indicated to Class I/II indications per guidelines/consensus released by Chinese Society of Cardiac Pacing and Electrophysiology
  2. Subject must have the ImageReady System as their initial (de novo) defibrillation system implant
  Interventions: Device: ImageReady™ MR Conditional Defibrillation System

INTERVENTIONS:
Device: ImageReady™ MR Conditional Defibrillation System — Subject will receive an ICD or CRT-D pulse generator in the left or right pectoral region ICD

SUMMARY:
To observe the safety and effectiveness of ImageReady™ MR conditional defibrillation system in a Chinese population.

DETAILED DESCRIPTION:
This is a multi-center, prospective, single-arm study, aimed to observe the safety and effectiveness of ImageReady™ MR conditional defibrillation system in a Chinese population.It will enroll 20 subjects in 5 sites in China.The primary safety endpoint is MR scan-related Complication-free rate between the MR Scan and the MRI + 1 Month Visit. The primary effectiveness endpoints include:1.Abnormal increase in RV shocking impedance from the pre-MR scan to the 1 Month post-MR scan. 2.Increase in RV pacing threshold from the pre-MR scan to the 1 Month post-MR scan. 3.Decrease in RV sensed amplitude from the pre-MR scan to the 1 Month post-MR scan. 4.Increase in LV pacing threshold from the pre-MR scan to the 1 Month post-MR scan. 5.Decrease in LV sensed amplitude from the pre-MR scan to the 1 Month post- MR scan.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is indicated to Class I/II indications per guidelines/consensus released by Chinese Society of Cardiac Pacing and Electrophysiology
2. Subject must have the ImageReady System as their initial (de novo) defibrillation system implant
3. Subject will receive an ICD or CRT-D pulse generator in the left or right pectoral region ICD
4. Subject is able and willing to undergo an MR scan
5. Subject is willing and capable of providing informed consent and participating in all testing/ visits associated with this clinical study at an approved clinical study center and at the intervals defined by this protocol
6. Subject is age 18 or above

Exclusion Criteria:

1. Subject has other active or abandoned implanted cardiac rhythm devices, components or accessories present such as pulse generators, leads, lead adaptors or extenders
2. Presence of metallic objects that represent a contraindication to MR imaging at the discretion of the Radiologist and impacting the ability to conduct the study protocol
3. Subject needs or will need a medically necessary MR scan, before completing the 1-month post-MR follow-up visit
4. Subject with:

   * A history of syncope related to brady-arrhythmia
   * A history of syncope of unknown etiology
   * Sinus pauses (Pause > 2 s)
   * Permanent or intermittent complete AV block
   * Documentation of progressive AV nodal block over time
   * Trifascicular block (alternating bundle branch block or PR > 200 ms with LBBB or other bifascicular block)

     * Note: It is required to run a 12 lead ECG and a 10s rhythm strip to document this exclusion criterion.
5. Subject is not clinically capable of tolerating the absence of pacing or Resynchronization therapy support in a supine position for the duration that the pulse generator is in MRI Protection Mode, per Physician discretion
6. Subject is not clinically capable of tolerating the absence of Tachycardia therapy support for the duration that the pulse generator is in MRI Protection Mode, per Physician discretion
7. Subjects currently requiring dialysis
8. Subject has a mechanical heart valve
9. Subject has a known or suspected sensitivity to dexamethasone acetate (DXA)
10. Subject is currently on the active heart transplant list
11. Subject has documented life expectancy of less than 12 months
12. Subject is enrolled in any other concurrent study that might interfere with this study
13. Women of childbearing potential who are or might be pregnant at the time of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yangang Su, Doctor, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nazarian S, Hansford R, Roguin A, Goldsher D, Zviman MM, Lardo AC, Caffo BS, Frick KD, Kraut MA, Kamel IR, Calkins H, Berger RD, Bluemke DA, Halperin HR. A prospective evaluation of a protocol for magnetic resonance imaging of patients with implanted cardiac devices. Ann Intern Med. 2011 Oct 4;155(7):415-24. doi: 10.7326/0003-4819-155-7-201110040-00004. PMID 21969340
- [Background] Russo RJ, Costa HS, Silva PD, Anderson JL, Arshad A, Biederman RW, Boyle NG, Frabizzio JV, Birgersdotter-Green U, Higgins SL, Lampert R, Machado CE, Martin ET, Rivard AL, Rubenstein JC, Schaerf RH, Schwartz JD, Shah DJ, Tomassoni GF, Tominaga GT, Tonkin AE, Uretsky S, Wolff SD. Assessing the Risks Associated with MRI in Patients with a Pacemaker or Defibrillator. N Engl J Med. 2017 Feb 23;376(8):755-764. doi: 10.1056/NEJMoa1603265. PMID 28225684
- [Background] ASTM Standard F2503-08, "Standard Practice for Marking Medical Devices and Other Items for Safety in the Magnetic Resonance Environment" ASTM International, West Conshohocken, PA, 2008, DOI: 10.1520/F2503-08, www.astm.org..
- [Background] Chinese Medical Association ECG Physiology and Pacing Branch, Chinese Medical Association Cardiology Branch, Chinese Medical Association Cardiology Professional Committee implanted cardioverter defibrillator treatment. Implanted cardioverter defibrillator treatment of China Expert consensus. Chinese Journal of Cardiac Arrhythmias 2014;18:242-53.
- [Background] Shu Zhang, Dejia Huang, Wei Hua, et al. Advice on cardiac resynchronization therapy for chronic heart failure (revised in 2013). Chinese Journal of Cardiac Arrhythmias 2013;17:247-61.
- [Background] Wolf SM, Lawrenz FP, Nelson CA, Kahn JP, Cho MK, Clayton EW, Fletcher JG, Georgieff MK, Hammerschmidt D, Hudson K, Illes J, Kapur V, Keane MA, Koenig BA, Leroy BS, McFarland EG, Paradise J, Parker LS, Terry SF, Van Ness B, Wilfond BS. Managing incidental findings in human subjects research: analysis and recommendations. J Law Med Ethics. 2008 Summer;36(2):219-48, 211. doi: 10.1111/j.1748-720X.2008.00266.x. PMID 18547191
- [Background] Kanal E, Barkovich AJ, Bell C, Borgstede JP, Bradley WG Jr, Froelich JW, Gilk T, Gimbel JR, Gosbee J, Kuhni-Kaminski E, Lester JW Jr, Nyenhuis J, Parag Y, Schaefer DJ, Sebek-Scoumis EA, Weinreb J, Zaremba LA, Wilcox P, Lucey L, Sass N; ACR Blue Ribbon Panel on MR Safety. ACR guidance document for safe MR practices: 2007. AJR Am J Roentgenol. 2007 Jun;188(6):1447-74. doi: 10.2214/AJR.06.1616. No abstract available. PMID 17515363

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was finished on 27Dec2018 and total 20 patients enrolled in study
Groups:
- ImageReady™ MR Conditional Defibrillation System: 1. Subject is indicated to Class I/II indications per guidelines/consensus released by Chinese Society of Cardiac Pacing and Electrophysiology
  2. Subject must have the ImageReady System as their initial (de novo) defibrillation system implant
  ImageReady™ MR Conditional Defibrillation System: Subject will receive an ICD or CRT-D pulse generator in the left or right pectoral region ICD
Period: Overall Study
Arm/Group | ImageReady™ MR Conditional Defibrillation System
Started | 20
Completed | 19
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | ImageReady™ MR Conditional Defibrillation System
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 7
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60.1 [26 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han Chinese | 20
Region of Enrollment [Count of Participants; unit: Participants]
  China | 20
Arrhythmia History [Count of Participants; unit: Participants]
  Atrioventricular block | 4
  Supraventricular Tachycardia | 1
  Atrial Fibrillation Paroxysmal | 2
  Atrial Fibrillation Persistent | 1
  Ventricular tachycardia / Ventricular Fibrillation | 9
  Other | 5
Cardiac Disease History [Count of Participants; unit: Participants]
  Hypertension | 11
  Diabetes | 5
  Renal Disease | 2
  Chronic Pulmonary Disease | 2
  Cerebrovascular Disease | 1
  Coronary Artery Disease (CAD) | 11
  Valvular Heart Disease | 3
  Heart Failure | 4
  Other | 11

OUTCOME MEASURES:

1. Primary Outcome: The Percent of Participants Who Were MR Scan-Related ImageReady System Complication -Free
Description: The primary safety endpoint of the MR ICD study will be assessed for all subjects who undergo any portion of the study-required MR scan sequences. Safety will be confirmed by evaluating the MR scan related ImageReady System complication-free rate (CFR) between the MR Scan and the MRI Visit + 1 Month.MR scan related ImageReady System complication is relation with ImageReady System and MR Scan.
Time Frame: MRI + 1 Month Visit（10-13 weeks from 0 day）
Population: 20 patients enrolled. 19 attended the MR scan.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ImageReady™ MR Conditional Defibrillation System
Number analyzed (Participants) | 19
percentage of participants | 100 [82.4 to 100]

2. Primary Outcome: The Percentage of Participant Whose the Average RV Shocking Impedance is >200 Ohm 1 Month Post Scan, While it is ≤ 200 Ohm Before Scan
Description: The normal RV shocking impedance measured by the system should be≤200 Ohm, with >200 Ohm considered abnormal. The primary effectiveness endpoint 1 is defined as that the average RV shocking impedance is >200 Ohm at 1 month post scan, while it is ≤ 200 Ohm before scan.There is no hypothesis testing in the MR ICD study, and it can be considered reasonable if up to 2 failed cases of primary effectiveness endpoint 1 occur.
Time Frame: MRI+1 Month visit ( 10~13 weeks from 0 day)
Population: 20 patients enrolled. 19 attended the MR scan.
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | ImageReady™ MR Conditional Defibrillation System
Number analyzed (Participants) | 19
percentage of participant | 0 [0 to 17.6]

3. Primary Outcome: The Percentage of Participant That Have an Increase in Average RV Pacing Thresholds > 0.5V (at 0.5 ms) From Pre-MR Scan to MRI Visit + 1 Month Follow-up
Description: Subjects that have an increase in average RV pacing thresholds ≤ 0.5V (at 0.5 ms) from pre-MR Scan to MRI Visit + 1 Month follow-up will be considered a success, otherwise, it is a primary effectiveness endpoint 2 event.The performance goal of this endpoint for the ENABLE MRI study was 87%. There is no hypothesis testing in the MR ICD study, and it can be considered reasonable if up to 2 failed cases of primary effectiveness endpoint 2 occur.
Time Frame: MRI+1Month visit( 10~14 weeks from 0 day)
Population: 20 patients enrolled.19 of them underwent the MR scan and the evaluation of RV pacing thresholds
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | ImageReady™ MR Conditional Defibrillation System
Number analyzed (Participants) | 19
percentage of participant | 0 [0 to 17.6]

4. Primary Outcome: The Percentage of Participant That Have the Average RV Sensed Amplitude at the MRI + 1 Month Visit Remains < 5.0 mV or Less Than 50% of the Pre-MR Scan Value
Description: Subjects will be considered a success if the average sensed amplitude at the MRI + 1 Month Visit remains ≥ 5.0 mV and above 50% of the pre-MR scan value, otherwise, it is a primary effectiveness endpoint 3 event.The performance goal of this endpoint for the ENABLE MRI study was 85%. There is no hypothesis testing in the MR ICD study, and it can be considered reasonable if up to 2 failed cases of primary effectiveness endpoint 3 occur.
Time Frame: MR+1 Month visit( 10~14 weeks from 0 day)
Population: 20 patients enrolled.19 of them underwent the MR scan and the evaluation of RV sensed amplitude
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | ImageReady™ MR Conditional Defibrillation System
Number analyzed (Participants) | 19
percentage of participant | 0 [0 to 17.6]

5. Primary Outcome: The Percentage of Participant Have an Increase in Average LV Pacing Thresholds >1.0V (at 0.5 ms) From Pre-MR Scan to MRI Visit + 1 Month Follow-up
Description: Subjects that have an increase in average LV pacing thresholds ≤1.0V (at 0.5 ms) from pre-MR Scan to MRI Visit + 1 Month follow-up will be considered a success, otherwise, it is a primary effectiveness endpoint 4 event.The performance goal of this endpoint for the ENABLE MRI study was 87%. There is no hypothesis testing in the MR ICD study, and it can be considered reasonable if up to 2 failed cases of primary effectiveness endpoint 4 occur.
Time Frame: MR +1 Month visit( 10~14 weeks from 0 day)
Population: only 10 patients implanted with LV leads and underwent the evaluation of LV pacing thresholds. Besides, 9 of them underwent the MR scan.
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | ImageReady™ MR Conditional Defibrillation System
Number analyzed (Participants) | 9
percentage of participant | 0 [0 to 33.6]

6. Primary Outcome: the Percentage of Participant That Have the Average LV Sensed Amplitude at the MRI + 1 Month Visit Remains <5.0 mV or Above 50% of the Pre-MR Scan Value
Description: Subjects will be considered a success if the average sensed amplitude at the MRI + 1 Month Visit remains ≥ 5.0 mV and above 50% of the pre-MR scan value, otherwise, it is a primary effectiveness endpoint 5 event.The performance goal of this endpoint for the ENABLE MRI study was 85%. There is no hypothesis testing in the MR ICD study, and it can be considered reasonable if up to 2 failed cases of primary effectiveness endpoint 5 occur.
Time Frame: MR +1 Month visit( 10~14 weeks from 0 day)
Population: only 10 patients implanted with LV leads and underwent the evaluation of LV sensed amplitude. Besides, 9 of them underwent the MR scan.
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | ImageReady™ MR Conditional Defibrillation System
Number analyzed (Participants) | 9
percentage of participant | 0 [0 to 33.6]

ADVERSE EVENTS:
Time Frame: Adverse event data were monitored at points of Enrollment, Implant, Pre-discharge, MRI Visit and MRI+1 Month visit.
Arm/Group | ImageReady™ MR Conditional Defibrillation System
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 6/20
Other Adverse Events (participants affected / at risk) | 11/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ImageReady™ MR Conditional Defibrillation System (N=20)
Cardiac failure congestive (Cardiac disorders) | 1 (2)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ImageReady™ MR Conditional Defibrillation System (N=20)
Cardiac failure acute (Cardiac disorders) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Implant site extravasation (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1)
Micturition disorder (Renal and urinary disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2)
Varicose vein (Vascular disorders) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Acid base balance abnormal (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Diaphragmatic spasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1)
Device stimulation issue (Product Issues) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT03451721/Prot_SAP_000.pdf